CLINICAL TRIAL: NCT03603197
Title: A Randomized, Double Blind and Placebo Controlled Multicenter Study Comparing BP-C1 and an Equal Looking Placebo in Metastatic Breast Cancer Patients. A Phase IIB Study
Brief Title: BP-C1 in Short-term Treatment of Thai Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meabco A/S (Industry)
Collaborators: Meddoc (Other); Norwegian University of Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MBC-BPC1/IIB
Record Dates: First submitted 2018-07-17; First posted 2018-07-27 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Breast Cancer; Stage IV Breast Cancer
Keywords: BP-C1; cis-coordinated complexes of platinum(II) with polymer of benzene polycarboxylic acids derived from lignin; Benzene polycarboxylic acids complex with cis-diammineplatinum(II); Metastatic Breast Cancer; Platinum analogue; Metronomic chemotherapy; Breast cancer; Cisplatin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BP-C1 (Experimental): Patients allocated to BP-C1 arm will be treated for 32 consecutive days. Patients who respond to treatment and do not experience untolerated toxicity will be invited to participate in the BMC2011-02 study, where they are offered to continue treatment with BP-C1.
  Interventions: Drug: BP-C1
- Placebo (Placebo Comparator): Patients allocated to Placebo arm will be treated for 32 consecutive days. Thereafter the patients will cross over to 32-day treatment with BP-C1. Patients who respond to treatment and do not experience untolerated toxicity will be invited to participate in the BMC2011-02 study, where they are offered to continue treatment with BP-C1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BP-C1 — BP-C1, 0.05% solution for injection; doses: 0.035 mg/kg body weight (0.07 mL/kg) intramuscularly once daily for 32 consecutive days
  Other Names: Cis-coordinated complexes of platinum(II) with polymer of benzene polycarboxylic acids derived from lignin; Cis-diammineplatinum(II) complexed with a polymer containing benzene polycarboxylic acids derived from lignin
  Arms: BP-C1
Drug: Placebo — Placebo, solution for injection; doses: 0.07 mL/kg body weight intramuscularly once daily for 32 consecutive days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether BP-C1 is effective in the short-term treatment of metastatic breast cancer patients who have previously undergone at least three lines of chemotherapy.

DETAILED DESCRIPTION:
BP-C1, solution for injection 0.05%, is currently being developed for treatment of patients with metastatic breast cancer with palliative intent.

Active substance of the product, which is a novel platinum-containing anticancer agent developed for intramuscular administration, is а cis-diammineplatinum(II) complexed with a polymer containing benzene polycarboxylic acids derived from lignin.

The amphiphilic characteristics of the polymer have resulted in a product with clear and significantly altered and improved properties compared to other platinum analogues, e.g. cisplatin, carboplatin and oxaliplatin.

BP-C1 preserves antitumour activity of its predecessors (e.g. cisplatin and carboplatin), additionally offering the following advantages that ensure favourable outcome of treatment of metastatic breast cancer patients:

* injectable solution (intramuscular) does not cause injection site reactions; can be administered at home by a nurse or a patient;
* has an improved pharmacokinetic profile;
* demonstrates efficacy comparable to cisplatin and much higher than carboplatin (in-vitro; in-vivo data);
* exerts an additional immunomodulatory activity.

This study is a randomised, double-blind, placebo-controlled, multicentre, phase IIb study in Thai patients with metastatic breast cancer. The eligible patients will be allocated (1:1) to either BP-C1 arm or Placebo arm and treated once daily for 32 days. The patients allocated to Placebo arm will cross over to BP-C1 treatment for 32 days when progression of the cancer will be documented and latest after 32-day treatment with Placebo. After 32-day treatment with BP-C1 the patients are invited to continue open-label treatment under protocol BMC2011-02.

ELIGIBILITY:
Inclusion Criteria:

Female patients with histologically verified metastatic breast cancer (stage IV) with measurable metastases, between 18 and 80 years of age, who had undergone at least three lines of chemotherapy and had an expected survival time of at least 3 months.

Exclusion Criteria:

Patients fulfilling at least one of the following criteria will be excluded from participation in the study:

* Abnormal liver function classified as total bilirubin >34 μmol/L or ALAT > 3 times of the upper limit of normal (ULN). In case of metastases in the liver, the ALAT limit for exclusion is set to 5хULN.
* Abnormal kidney function defined by serum creatinine >120 μmol/L.
* Abnormal coagulation capacity defined by the relative arbitrary concentration of coagulation factors 2,7,10; INR >1.5.
* Verified metastases to the brain.
* Synchronous cancer except for non- melanoma skin cancer and early stage of cervical cancer.
* Abnormal hematology status defined by hemoglobin < 9.0 g/dL, platelet count < 100,000/mm^3 or leucocytes < 3 x 10^9/L.
* Clinically significant abnormal ECG.
* Karnofsky performance status score <60%.
* Pregnant or breast feeding women.
* Women of fertile age who do not want to be tested for possible pregnancy.
* Fertile female who do not want to use safe protection against pregnancy, starting one month before the start of the study treatment and lasting at least six weeks after.
* Uncontrolled bacterial, viral, fungal or parasite infection.
* Under systemic treatment with corticosteroids or other immunosuppressive drugs in the last 21 days before start of the trial treatment.
* Participating in another clinical trial with pharmaceuticals in the last six weeks before start of this trial treatment.
* Not able to understand information.
* Not willing or not able to give written consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Change (%) in the sum of diameters of target lesions | baseline to Day 32 of treatment
  Diameter of target lesions will be measured by computer tomography (CT) with contrasting using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Number of target lesions | baseline to Day 32 of treatment
  Number of target lesions per each patient will be evaluated by CT with contrasting. Number of target lesions at baseline and Day 32 of treatment will be presented in shift tables.
Treatment response | baseline to Day 32 of treatment
  In accordance with RECIST v1.1 the treatment response will be classified as 'complete response', 'partial response', 'stable disease' or 'progressive disease':
  Complete response (CR): disappearance of all target lesions. Partial response (PR): at least 30% decrease in the sum of longest diameters of target lesions, taking as reference the baseline sum of diameters.
  Progressive disease (PD): at least 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum might also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions will also be considered progression.
  Stable disease (SD): neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Karnofsky Performance Status (KPS) score | baseline to Day 16 and Day 32 of treatment
  KPS describes an outcome in 11 grades, starting as normal without complaints and evidence of disease (equals 100 as the best) and dead (equals 0) as the lowest. KPS score will be assessed every 16 days during 32-day treatment period.
Separate scores of the general questionnaire EORTC QLQ-C30 | baseline to Day 16 and Day 32 of treatment
  The EORTC QLQ-C30 is a general quality of life questionnaire for cancer patients. The questionnaire contains 30 questions. Three variables will be obtained from the EORTC QLQ-C30: the sum of scores C1 to C5 denoted as "Physical activity problem last week", the sum of scores C6 to C28 denoted as "Discomfort last week", and the sum of scores C29 and C30 denoted as "Health and quality of life".
Separate scores of the specific questionnaire EORTC QLQ-BR23 | baseline to Day 16 and Day 32 of treatment
  The EORTC QLQ-BR23 is a breast cancer-specific quality of life questionnaire. The questionnaire consists of 23 questions. Three variables will be obtained from the EORTC-BR23: the sum of scores BR1 to BR13 denoted as "Breast cancer problem last week", the sum of scores BR14 to BR16 denoted as "Sexual interest and activity last four weeks" and the sum of scores BR17 to BR23 denoted as "Breast cancer related pain and discomfort last week".
Maximum Common Toxicity Criteria (CTC) score | baseline to Day 16 and Day 32 of treatment
  Maximum CTC score will be recorded using NCI Common Toxicity Criteria v2.0 divided in 15 categories.
Change in the Sum CTC score | baseline to Day 16 and Day 32 of treatment
  The Sum CTC score will be a sum of all registered CTC scores by 15 categories.
Number of registered adverse events | baseline to Day 32 of treatment
  Adverse events (AEs) will be coded according to the MedDRA (version 16.1E). AEs will be systemized by system organ class and by preferred term. AEs will be analyzed by severity, seriousness and relatedness to the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Kritiya Butthongkomvong, MD, Principal Investigator — Udon Thani Cancer Hospital, Thailand
Locations (4):
- Thailand (4):
  - Udon Thani Cancer Hospital, Udon Thani, Changwat Udon Thani
  - Siriraj Hospital, Mahidol University, Bangkok
  - Lampang Cancer Center, Lampang
  - Ubon Ratchanthani Cancer Hospital, Ubon Ratchathani

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Butthongkomvong K, Raunroadroong N, Sorrarichingchai S, Sangsaikae I, Srimuninnimit V, Harling H, Larsen S. Efficacy and tolerability of BP-C1 in metastatic breast cancer: a Phase II, randomized, double-blind, and placebo-controlled Thai multi-center study. Breast Cancer (Dove Med Press). 2019 Jan 14;11:43-51. doi: 10.2147/BCTT.S174298. eCollection 2019. PMID 30666153
- See also: Efficacy and tolerability of BP-C1 in metastatic breast cancer: a Phase II, randomized, double-blind, and placebo-controlled Thai multi-center study. — http://www.ncbi.nlm.nih.gov/pubmed/30666153